CLINICAL TRIAL: NCT05533268
Title: Efficacy of Mental and Physical Training on Blood Pressure and Resting Heart Rate Among Physically Inactive Young Adults With Elevated and High Blood Pressure
Brief Title: Effect of Mental and Physical Training on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MAP vs DASH Diet
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Elevated Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Physical Conditioning, Human; Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will not know about grouping of the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mental Training (Experimental): mindfulness meditation for 6-weeks.
  Interventions: Other: Mental training
- Physical Training (Experimental): Continuous moderate-intensity training for 6-weeks.
  Interventions: Other: Physical training
- Mental and Physical Training (Experimental): Combination of mindfulness meditation and continuous moderate-intensity training for 6 weeks.
  Interventions: Other: Mental & physical training
- DASH Diet Plan (Active Comparator): Dietary Approaches to Stop Hypertension for 6-weeks.
  Interventions: Other: DASH diet

INTERVENTIONS:
Other: Mental training — Mental training (guided mindfulness meditation by Jon Kabat-Zinn for 20 minutes, 3 times per week.
  Arms: Mental Training
Other: Physical training — Physical training (continuous moderate-intensity training at 40-60% of participants' heart rate reserve for 20 minutes excluding warm-up/cool-down, 3 times per week.
  Arms: Physical Training
Other: Mental & physical training — Mental and physical training (combination of mindfulness mediation for 20-minutes, 3 times per week and continuous moderate-intensity training for 20 minutes, 3 times per week.
  Arms: Mental and Physical Training
Other: DASH diet — DASH diet ( (more vegetables, fruits and low-fat dairy foods and moderate amounts of whole grains, fish, poultry and nuts; and less than 3 grams of sodium daily) for 6-weeks.
  Arms: DASH Diet Plan

SUMMARY:
Elevated blood pressure or prehypertension is highly associated with increased risk of developing hypertension, cardiovascular event, and type II diabetes. Many physically inactive young adults, particularly in Malaysia have blood pressure higher than normal range, therefore it is important to control the blood pressure within normal range as prophylactic measure. This experimental research will be carried out to study the effect of physical training (aerobic exercise) and mental training (mindfulness meditation) with diet as a control group on the systolic blood pressure, diastolic blood pressure and resting heart rate among young adult with elevated blood pressure living a sedentary lifestyle. Participant will be divided into 2 experimental groups (mental and physical training) and 1 control group (Dietary Approaches to Stop Hypertension -DASH diet plan) who need to complete the prescribed intervention for 6 weeks. Results will be analysed by repeated measures ANOVA followed by post-hic test.

ELIGIBILITY:
Inclusion Criteria:

* Male adults aged 18-25 years
* Normal BMI (18.5-24.9)
* Physically inactive
* SBP between 120-139 mmHg and/or DBP between 60-89 mmHg
* No hearing abnormalities
* Willing to participate

Exclusion Criteria:

* Participants who have cardiovascular, musculoskeletal, and neurological disorders or any other medical condition that would restrict them to participate in the exercise
* Those who are taking antihypertensive medications or other medications that will affect their BP and heart rate
* Participants who are currently engaging in any form of relaxation techniques such as yoga or meditation
* Individuals who are actively engaged in physical activities

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Young male adults who are physically inactive.
Enrollment: 62 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure at 6 weeks. | At baseline over a period of 6 weeks.
  Systolic blood pressure (SPB) will be measured at baseline (before intervention begin), after 3 weeks of intervention, and post 6-weeks of intervention.
Change from Baseline Diastolic Blood Pressure at 6 weeks. | At baseline over a period of 6 weeks.
  Diastolic blood pressure (DPB) will be measured at baseline (before intervention begin), after 3 weeks of intervention, and post 6-weeks of intervention.
Change from Baseline Mean Arterial Pressure at 6 weeks. | At baseline over a period of 6 weeks.
  Mean arterial pressure (MAP) will be measured at baseline (before intervention begin), after 3 weeks of intervention, and post 6-weeks of intervention.
Change from Baseline Resting Heart Rate at 6 weeks. | At baseline over a period of 6 weeks.
  Resting heart rate (RHR) will be measured at baseline (before intervention begin), after 3 weeks of intervention, and post 6-weeks of intervention.
Change from Baseline Pulse Pressure at 6 weeks. | At baseline over a period of 6 weeks.
  Pulse pressure will be measured at baseline (before intervention begin), after 3 weeks of intervention, and post 6-weeks of intervention.

SECONDARY OUTCOMES:
Change from Baseline Body Mass Index at 6 weeks. | At baseline over a period of 6 weeks.
  Body mass index (BMI) will be measured at baseline (before intervention begin), after 3 weeks of intervention, and post 6-weeks of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
IDP will not be shared.